CLINICAL TRIAL: NCT04028193
Title: The Effect of Fat Supplementation on the Appearance of Symptoms Associated With Dumping Syndrome in Patients Undergone Bariatric Surgery
Brief Title: Fat Supplementation on Dumping Syndrome Associated Symptoms
Acronym: Fat on DS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technological Educational Institute of Thessaly (Other)
Responsible Party: Principal Investigator, Chatzipapa Nikoleta, Research Associate University of Thessaly, University of Thessaly
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5411069DD0467
Record Dates: First submitted 2019-07-15; First posted 2019-07-22 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Dumping Syndrome
Keywords: Dumping syndrome; Fat supplement; post bariatric surgery
MeSH Terms: conditions — Dumping Syndrome | interventions — Energy-Generating Resources

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diagnose Dumping after supplement consumption (Other): Carbohydrate ingestion to provoke dumping syndrome related symptoms
  Interventions: Dietary Supplement: Resource Energy
- Fat supplementation (Other): A high fat supplement was added to the carbohydrate liquid meal that was previously used for diagnosis.
  Interventions: Dietary Supplement: Calogen

INTERVENTIONS:
Dietary Supplement: Calogen — Polyunsaturated liquid fat supplement
  Other Names: Calogen fat supplement
  Arms: Fat supplementation
Dietary Supplement: Resource Energy — Carbohydrate Supplement
  Arms: Diagnose Dumping after supplement consumption

SUMMARY:
The purpose of the study is the investigation of the effect of fat supplement on gastric emptying rate and the appearance of symptoms of Dumping Syndrome in patients who have undergone gastrointestinal- duodenal surgery. Patients who have undergone bariatric surgery have been examined for the presence of the Dumping syndrome, with glucose measurements, the Sigstad's questionnaire and questionnaire of Arts. Patients diagnosed positive, reiterated the examination process in a second meeting consuming an extra fat supplement. The data obtained on the different appointments were compared between the two groups in a cross over design.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Dumping Syndrome

Exclusion Criteria:

* Patients with diabetes mellitus type 1 and 2, Patients with impaired balance of fluids and electrolytes, Patients on diuretics pills or corticosteroids or hypoglycemic tablets and Insulin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Glucose Levels | before the ingestion of the carbohydrate and fat supplement (baseline)
  Blood glucose measurement
Glucose Levels | 30 minutes after the ingestion of the carbohydrate and fat supplement
  Blood glucose measurement
Glucose Levels | 60 minutes after the ingestion of the the carbohydrate and fat supplement
  Blood glucose measurement
Glucose Levels | 90 minutes after the ingestion of the the carbohydrate and fat supplement
  Blood glucose measurement
Glucose Levels | 120 minutes after the ingestion of the the carbohydrate and fat supplement
  Blood glucose measurement
Sigstad's Questionnaire | 1st hour after the ingestion of the supplements
  Dumping syndrome symptom associated questionnaire
Sigstad's Questionnaire | 2nd hour after the ingestion of the supplements
  Dumping syndrome symptom associated questionnaire
Arts's Questionnaire | 1st hour after the ingestion of the supplements
  Dumping syndrome symptom associated questionnaire
Arts's Questionnaire | 2nd hour after the ingestion of the supplements
  Dumping syndrome symptom associated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Nikoleta Chatzipapa, Thessaloniki, Greece